CLINICAL TRIAL: NCT02797938
Title: Comparison of the Endotracheal Tube Cuff Pressure Between a Taper-guard Cuffed Tube and a Cylindrical-shaped Cuffed Tube After Changing in Position During Middle Ear Surgery
Brief Title: Comparison of the Cuff Pressure Between a Taper-guard Cuffed Tube and a Cylindrical-shaped Cuffed Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KNUH 2016-02-017-001
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cuff Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taper guard tube (Experimental): Taper guard tube was intubated in 26 patients
  Interventions: Device: Taper guard tube
- Cylindrical tube (Active Comparator): Cylindrical tube was intubated in 26 patients
  Interventions: Device: Cylindrical tube

INTERVENTIONS:
Device: Taper guard tube — Taper guard tube was intubated
  Arms: Taper guard tube
Device: Cylindrical tube — Cylindrical tube was intubated
  Arms: Cylindrical tube

SUMMARY:
Endotracheal pressure with different cuff shapes can result in different cuff pressure change after head positional change. In this study, 52 patients underwent middle ear surgery with general anesthesia were randomly allocated to two group; patients were intubated with taper guard cuffed tube or cylindrical shaped cuffed tube. Anesthesia was maintained with sevoflurane with air/oxygen and remifentanil. The cuff pressure was initially set at 22 centimeters of water in the neural head position and was measured after the change to the 45 degree head rotation. The change of cuff pressure was compared between two groups

DETAILED DESCRIPTION:
Endotracheal pressure with different cuff shapes can result in different cuff pressure change after head positional change. In this study, 52 patients underwent middle ear surgery with general anesthesia were randomly allocated to two group; patients were intubated with taper guard cuffed tube or cylindrical shaped cuffed tube. Anesthesia was maintained with sevoflurane with air/O2 and remifentanil. The cuff pressure was initially set at 24 centimeters of water in the neural head position and was measured after the change to the 45 degree head rotation. In addition, sore throat, hoarseness , dysphagia and cough were recorded 0, 6, 12, 24 hr after surgery. The change of cuff pressure was compared between two groups. The side effects associated with tube were compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent middle ear surgery with general anesthesia American Society of Anesthesiology status 1-3

Exclusion Criteria:

* Patient with neck pain Patient with a history of neck surgery Patient with limited movement of neck Patient with body mass index more than 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change of cuff pressure | 5 minutes after rotation of 45 degree of head
  Change of cuff pressure of endotracheal tube after rotation 45 degree of head

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes